CLINICAL TRIAL: NCT03538782
Title: Retrospective Multicenter Study on Patients Radiation Exposure in Percutaneous Transhepatic Biliary Drainage (PTBD) Procedures.
Brief Title: Patients Radiation Exposure in Percutaneous Transhepatic Biliary Drainage (PTBD) Procedures
Status: Completed | Type: Observational
Sponsor: Theresienkrankenhaus und St. Hedwig-Klinik GmbH (Other)
Collaborators: The Federal Office for Radiation Protection, Germany (Other Government)
Responsible Party: Principal Investigator, Daniel Schmitz, Principal investigator, Theresienkrankenhaus und St. Hedwig-Klinik GmbH
Other Study IDs: Rad Exp PTBD 2018 V1.0
Record Dates: First submitted 2018-05-12; First posted 2018-05-29 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Radiation Exposure
Keywords: percutaneous biliary drainage; radiation exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous biliary drainage — The initial puncture of the bile duct with an access needle is performed by ultrasound guidance or by fluoroscopic guidance. After injection of the radiopaque contrast media into the bile duct system the rest of the examination is performed by fluoroscopic guidance. All different PTBD procedures are analyzed: insertion, exchange or removal of a plastic catheter, metal stent implantation, PTBD with cholangioscopy, PTBD with ballon dilatation, PTBD with lithotrypsy or diagnostic percutaneous transhepatic cholangiography.

SUMMARY:
Percutaneous transhepatic biliary drainage (PTBD) procedures are associated with an elevated radiation exposure for the patient. In the recently published guideline of the Federal Ofﬁce for Radiation Protection in Germany diagnostic reference levels (DRLs) for dose area products (DAP) are not defined for PTBD procedures due to insufficient data. The aim of this retrospective study is to give a nation-wide survey on patients radiation exposure in different PTBD procedures considering factors that may have an impact on increased radiation exposure like fluoroscopic-guided versus ultrasound-guided bile duct puncture.

DETAILED DESCRIPTION:
Percutaneous transhepatic biliary drainage (PTBD) procedures are associated with an elevated radiation exposure for the patient. Usually, radiation exposure in radiological interventions is measured by the dose area product (DAP). Diagnostic reference levels (DRLs) are based on the third quartiles (Q3) of the pooled dose area product (DAP) for the known interventional procedures. They have been introduced in the 1980s by the International Commission on Radiological Protection's (ICRP's) to reduce patients radiation exposure. In the recently published guideline of the Federal Ofﬁce for Radiation Protection in Germany in 2016 DRLs are not defined for PTBD procedures due to insufficient data. Procedure complexity due to different techniques, patient anatomy, lesion characteristics and disease severity makes it difficult to define DRLs in this fluoroscopy-guided intervention. The ICRP recently published some recommendations on DRLs in medical imaging including radiological interventions. As DRLs are often missing in this field, it was suggested to analyze national data sets comprising dosimetric data from a large number of facilities. The aim of this retrospective study is to give a nation-wide survey on patients radiation exposure in different PTBD procedures considering factors that may have an impact on increased or decreased radiation exposure like fluoroscopic-guided versus ultrasound-guided bile duct puncture. A questionnaire was sent to 200 gastroenterological and radiological departments in university and non-university hospitals to analyze the last 10 - 30 consecutively performed PTBD procedures.

ELIGIBILITY:
Inclusion Criteria:

* 10 up to 30 consecutively performed PTBDs are documented in the study center
* body weight of the examined patients is about 60 - 80 kilogramms
* returned questionaire is complete in regard to DAP, fluoroscopy time, number of still images, characters of the intervention, characterization of the fluoroscopy device (manufacturer, date of first registration)

Exclusion Criteria:

* the study center performs less than 10 PTBDs/year
* returned questionaire is incomplete

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutively performed PTBDs in each study center are included taking account of the exclusion/inclusion criteria
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Radiation Exposure | From the beginning of the radiological examination until the end the examination (15 - 180 minutes)
  Radiation Exposure for the patient is measured by the dose area product (cGy x cm2 resp.µGy x∙m2)

SECONDARY OUTCOMES:
Fluoroscopy time | From the beginning of the radiological examination until the end the examination (15 - 180 minutes)
  Accumulated fluoroscopy time for the complete examination (minutes)
Number of images | From the beginning of the radiological examination until the end the examination (15 -180 minutes)
  Number of still images which are produced during the whole examination (n)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Schegerer, Dr.rer.nat., Study Director — Federal Office of Radiation Protection, Germany
Locations (1):
- Universitätsklinikum des Saarlandes und Medizinische Fakultät der Universität des Saarlandes Klinik für Innere Medizin II - Gastroenterologie und Endokrinologie, Bad Homburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kloeckner R, Bersch A, dos Santos DP, Schneider J, Duber C, Pitton MB. Radiation exposure in nonvascular fluoroscopy-guided interventional procedures. Cardiovasc Intervent Radiol. 2012 Jun;35(3):613-20. doi: 10.1007/s00270-011-0206-y. Epub 2011 Jul 27. PMID 21792735
- [Background] Stratakis J, Damilakis J, Hatzidakis A, Perisinakis K, Gourtsoyiannis N. Radiation dose and risk from fluoroscopically guided percutaneous transhepatic biliary procedures. J Vasc Interv Radiol. 2006 Jan;17(1):77-84. doi: 10.1097/01.RVI.0000188754.97465.13. PMID 16415136
- [Background] Ruiz-Cruces R, Vano E, Carrera-Magarino F, Moreno-Rodriguez F, Soler-Cantos MM, Canis-Lopez M, Hernandez-Armas J, Diaz-Romero FJ, Rosales-Espizua F, Fernandez-Soto JM, Sanchez-Casanueva R, Martin-Palanca A, Perez-Martinez M, Gil-Agudo A, Zarca-Diaz MA, Parra-Osorio V, Munoz Ruiz-Canela JJ, Moreno-Sanchez T, Lopez-Medina A, Moreno-Saiz C, Galan-Montenegro P, Gallego-Beuter JJ, Gonzalez-de-Garay M, Zapata-Jimenez JC, Pastor-Vega JM, Canete S. Diagnostic reference levels and complexity indices in interventional radiology: a national programme. Eur Radiol. 2016 Dec;26(12):4268-4276. doi: 10.1007/s00330-016-4334-2. Epub 2016 Jul 6. PMID 27384609
- See also: Diagnostic Reference Levels in Medical Imaging ICRP Publication 135 — http://www.icrp.org/publication.asp?id=ICRPPublication135
- See also: Bekanntmachung der aktualisierten diagnostischen Referenzwerte für diagnostische und interventionelle Röntgenanwendungen 2016 — http://www.bfs.de/DE/themen/ion/anwendung-medizin/diagnostik/referenzwerte/referenzwerte_node.html